CLINICAL TRIAL: NCT01932554
Title: Abciximab (ReoPro) as a Therapeutic Intervention for Sickle Cell Vaso-Occlusive Pain Crisis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: St. Louis University (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Principal Investigator, William Ferguson M.D., Professor of Pediatrics, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SLU 23331
Record Dates: First submitted 2013-08-19; First posted 2013-08-30 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Sickle Cell Disease; Hb-SS Disease With Vasoocclusive Pain; Hemoglobin SS Disease With Vasoocclusive Crisis; Other Sickle Cell Disease With Vaso-Occlusive Pain; Hemoglobin SS Disease With Crisis
Keywords: Sickle Cell Pain Crisis; Abciximab; Integrins; Cell Adhesion Molecules
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Abciximab; Ibuprofen; Morphine; Hydromorphone; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abciximab (Experimental): Abciximab will be administered as initial bolus of dose of 0.25 mg/kg, delivered via syringe pump over 15 minutes, followed by a continuous infusion of 0.125 microgram/kg/min (max of 10 micrograms/min) infused over the next 12 hours. Infusion to start within 16 hours of admission.
  Patients will receive standard supportive care, including intravenous hydration, supplemental oxygen, incentive spirometry, ibuprofen, and parenteral narcotic pain medications (morphine, hydromorphone or fentanyl)
  Interventions: Drug: Abciximab; Other: Intravenous hydration; Drug: Ibuprofen; Drug: Parenteral narcotic; Other: Incentive spirometry; Other: Supplemental oxygen
- Placebo (Placebo Comparator): Inactive placebo will be administered as initial bolus followed by a continuous infusion over the next 12 hours, in syringes and volumes identical with the drug administered in the experimental arm. Infusion to begin within 16 hours of admission.
  Patients will receive standard supportive care, including intravenous hydration, supplemental oxygen, incentive spirometry, ibuprofen, and parenteral narcotic pain medications (morphine, hydromorphone or fentanyl)
  Interventions: Drug: Placebo; Other: Intravenous hydration; Drug: Ibuprofen; Drug: Parenteral narcotic; Other: Incentive spirometry; Other: Supplemental oxygen

INTERVENTIONS:
Drug: Abciximab — Abciximab will be administered as initial bolus of dose of 0.25 mg/kg, delivered via syringe pump over 15 minutes, followed by a continuous infusion of 0.125 microgram/kg/min (max of 10 micrograms/min) infused over the next 12 hours. Infusion to start within 16 hours of admission. All patients will receive standard supportive care measures.
  Other Names: ReoPro
  Arms: Abciximab
Drug: Placebo — Inactive placebo will be administered as initial bolus followed by a continuous infusion over the next 12 hours, in syringes and volumes identical with the drug administered in the experimental arm. Infusion to begin within 16 hours of admission. All patients will also receive standard supportive care measures.
  Arms: Placebo
Other: Intravenous hydration — intravenous hydration to provide total fluid intake of 1.25-1.5 times maintenance fluid requirements
Drug: Ibuprofen — Scheduled ibuprofen,~10 mg/kg every 6-8 hours
  Other Names: Advil, Motrin
Drug: Parenteral narcotic — Parenteral morphine administered by bolus or patient-controlled analgesia to maintain pain control. Hydromorphone or fentanyl will be used in patients who do not tolerate morphine.
  Other Names: morphine; hydromorphone; Dilaudid; fentanyl
Other: Incentive spirometry — Patients will perform incentive spirometry every 2 hours while awake
Other: Supplemental oxygen — Supplemental oxygen by nasal cannula or mask will be provided if needed to maintain oxygen saturation of 92% or greater.

SUMMARY:
The purpose of this study is to determine whether giving abciximab (ReoPro) to children with sickle cell disease who are hospitalized for acute pain crisis will improve their pain and shorten the time spent in the hospital, when compared with standard supportive care.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is one of the more common genetic diseases worldwide, affecting approximately 1 in 500 African-Americans and 1 in 1000 Hispanic-Americans. A single amino acid substitution decreases the solubility of deoxygenated hemoglobin, leading to polymer formation and subsequent distortion of erythrocyte shape from the normal biconcave disc into a relatively rigid crescent or sickle shape. Initially reversible, the polymer formation and shape distortion eventually becomes permanent. Clinical manifestations of sickle cell disease relate both to increased clearance of these misshapen erythrocytes (causing a chronic hemolytic anemia) as well as occlusion of small (and sometimes large) blood vessels.

Vaso-occlusive phenomena are responsible for much of the acute morbidity of sickle cell disease, including episodes of pain resulting from bone infarcts, splenic infarction with a secondary increased risk of infection, and a relatively high incidence of ischemic stroke (~10% in the first 2 decades of life). In addition, chronic and cumulative ischemic episodes contribute to long-term morbidity (including avascular necrosis of bone, retinopathy, renal insufficiency, and pulmonary hypertension) and a significantly shortened life span. Vaso-occlusive pain crises often require hospitalization for the administration of parenteral narcotics; the average duration of hospitalization is 4-5 days, and a significant proportion of patients experience multiple crises per year. In most episodes, pain continues to intensify over the first 2-3 days before beginning to abate, suggesting that there is ongoing extension of tissue damage for some time following initiation of the episode; also, many patients will develop additional foci of pain even during the course of hospitalization.

While direct mechanical blockage of small vessels by sickled erythrocytes is undoubtedly an important factor in vaso-occlusion, there are other secondary phenomena that are likely to contribute to these episodes, including increased erythrocyte adhesion to the endothelium of post-capillary venules. SCD patients also exhibit chronic pro-coagulation changes in soluble clotting factors, as well as increased platelet number and activation. The relative contribution of these various changes to the pathophysiology of vaso-occlusive crises is unclear. One published study showed that the antiplatelet drug ticlopidine decreased frequency, duration, and severity of pain crises in SCD patients, suggesting that the increase in platelet activation does indeed contribute to vaso-occlusion.

Current therapy for vaso-occlusive pain crises is mostly supportive (maintaining adequate hydration and oxygenation and administering pain medication). With the possible exception of exchange transfusion-a procedure with significant potential morbidity-there is no therapy that directly targets the vaso-occlusion.

Abciximab (ReoPro) is the Fab fragment of the chimeric human-mouse monoclonal antibody 7E3. It avidly binds to both glycoprotein IIb/IIIa and to integrin αvβ3, and so would potentially inhibit both erythrocyte binding to vascular endothelial as well as platelet adhesion, thus targeting two separate mechanisms that are felt to be components of the vaso-occlusive phenomenon in SCD.

The relatively prolonged course of most pain crises-which typically involves increasing intensity of pain and often development of new areas of pain over the first few days-suggests that treatment during the early phases of a crisis might be effective in ameliorating the course of the episode, resulting not only in decreased acute morbidity but possibly also in less long-term tissue damage. The study hypothesis is that administration of abciximab early in the course of a vaso-occlusive sickle cell pain crisis will reduce the median length of hospitalization without an accompanying increase in bleeding or other serious complications.

Participants will be randomized in a double blind fashion to receive either abciximab (ReoPro) or placebo intravenously over 12 hours. Randomization will be stratified by sickle cell genotype: Sickle Cell Anemia (SS) vs. Sickle-Hemoglobin C Disease (SC). All patients will receive standard supportive care, including hydration, supplemental oxygen as needed to maintain oxygen saturation >92%, scheduled use of NSAIDS, and narcotics titrated to effect.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of sickle cell disease (Hb SS, HbSC, HbS-β0-thalassemia)
2. Age 5.00 to 24.99 years
3. Pain consistent with vaso-occlusive crisis that meets the criteria for hospitalization and parenteral narcotics: moderate-severe pain unresponsive to oral medications (NSAIDS + narcotics) that has no alternative etiology (e.g., trauma)
4. Platelet count >100,000
5. INR <1.2, PTT < 40 seconds
6. Negative urine pregnancy test for females of child-bearing potential, including any female ≥10 years of age
7. Informed consent by patient (≥18 years of age) or parent (if patient <18 years of age); assent from patients 12-18 years of age
8. Ability to start drug/placebo infusion within 16 hours of admission

Exclusion Criteria:

1. History of stroke (either ischemic or hemorrhagic)
2. Currently receiving anticoagulation medication (heparin within 1 week, Coumadin within 3 weeks) or medication with irreversible anti-platelet effect (e.g., aspirin, ticlopidine) within 14 days
3. Red cell transfusion within 60 days
4. Major surgery within 30 days
5. Treatment with hydroxyurea within 30 days (due to evidence that hydroxyurea can reverse platelet activation in patients with SCD)
6. Tmax ≥ 102.0o F without concomitant signs of infection, or ≥ 100.4o F with any finding suggestive of bacterial infection, including acute chest syndrome (fever, respiratory symptoms, and new infiltrate on chest X-ray)
7. Active internal bleeding
8. Known allergy to abciximab or murine proteins
9. Recent (within 6 weeks) gastrointestinal or genitourinary bleeding of clinical significance
10. Bleeding diathesis
11. History of vasculitis
12. Intracranial neoplasm, arteriovenous malformation or aneurysm
13. Severe uncontrolled hypertension
14. Patients who previously participated in the study must be excluded due to the increased risk of severe thrombocytopenia.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalization | Duration of hospital stay, expected average of 5 days
  Total duration from admission to the inpatient service until discharge order is written, measured in days.

SECONDARY OUTCOMES:
Total narcotic dose | Duration of hospital stay, expected average of 5 days
  Total dose of parenteral narcotic administered during hospitalization, expressed as morphine equivalent per kg, will be calculated.
Bleeding complications | From randomization until 10 days following initial discharge from hospital
  All major or minor bleeding manifestations during hospitalization or in the immediate post-discharge period, including site and severity, will be tracked
Complications (other than bleeding) attributed to study drug | From randomization until 3 months following initial discharge from hospital
  All complications potentially related to abciximab therapy, other than bleeding, will be tracked.
Readmission rate | From discharge date until 3 months following initial discharge from hospital
  All readmissions for any cause occurring within 3 months of discharge will be tracked.

CONTACTS AND LOCATIONS:
Overall Officials: William S Ferguson, MD, Principal Investigator — St. Louis University
Locations (1):
- Cardinal Glennon Children's Medical Center, St Louis, Missouri, United States

REFERENCES:
- [Background] Dean J, Schechter AN. Sickle-cell anemia: molecular and cellular bases of therapeutic approaches (first of three parts). N Engl J Med. 1978 Oct 5;299(14):752-63. doi: 10.1056/NEJM197810052991405. No abstract available. PMID 357967
- [Background] Dean J, Schechter AN. Sickle-cell anemia: molecular and cellular bases of therapeutic approaches (second of three parts). N Engl J Med. 1978 Oct 12;299(15):804-11. doi: 10.1056/NEJM197810122991504. No abstract available. PMID 692564
- [Background] Bunn HF. Pathogenesis and treatment of sickle cell disease. N Engl J Med. 1997 Sep 11;337(11):762-9. doi: 10.1056/NEJM199709113371107. No abstract available. PMID 9287233
- [Background] Lane PA. Sickle cell disease. Pediatr Clin North Am. 1996 Jun;43(3):639-64. doi: 10.1016/s0031-3955(05)70426-0. PMID 8649903
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Steinberg MH. Management of sickle cell disease. N Engl J Med. 1999 Apr 1;340(13):1021-30. doi: 10.1056/NEJM199904013401307. No abstract available. PMID 10099145
- [Background] Rees DC, Olujohungbe AD, Parker NE, Stephens AD, Telfer P, Wright J; British Committee for Standards in Haematology General Haematology Task Force by the Sickle Cell Working Party. Guidelines for the management of the acute painful crisis in sickle cell disease. Br J Haematol. 2003 Mar;120(5):744-52. doi: 10.1046/j.1365-2141.2003.04193.x. No abstract available. PMID 12614204
- [Background] Hebbel RP. Perspectives series: cell adhesion in vascular biology. Adhesive interactions of sickle erythrocytes with endothelium. J Clin Invest. 1997 Jun 1;99(11):2561-4. doi: 10.1172/JCI119442. No abstract available. PMID 9169483
- [Background] Kaul DK, Tsai HM, Liu XD, Nakada MT, Nagel RL, Coller BS. Monoclonal antibodies to alphaVbeta3 (7E3 and LM609) inhibit sickle red blood cell-endothelium interactions induced by platelet-activating factor. Blood. 2000 Jan 15;95(2):368-74. PMID 10627437
- [Background] Finnegan EM, Barabino GA, Liu XD, Chang HY, Jonczyk A, Kaul DK. Small-molecule cyclic alpha V beta 3 antagonists inhibit sickle red cell adhesion to vascular endothelium and vasoocclusion. Am J Physiol Heart Circ Physiol. 2007 Aug;293(2):H1038-45. doi: 10.1152/ajpheart.01054.2006. Epub 2007 May 4. PMID 17483236
- [Background] Ataga KI, Orringer EP. Hypercoagulability in sickle cell disease: a curious paradox. Am J Med. 2003 Dec 15;115(9):721-8. doi: 10.1016/j.amjmed.2003.07.011. PMID 14693325
- [Background] Ataga KI, Key NS. Hypercoagulability in sickle cell disease: new approaches to an old problem. Hematology Am Soc Hematol Educ Program. 2007:91-6. doi: 10.1182/asheducation-2007.1.91. PMID 18024615